CLINICAL TRIAL: NCT03881670
Title: On-Eye Optical Quality of Lotrafilcon B Lenses Over 12 Hours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Pete Kollbaum, OD, PhD, Associate Professor, Associate Dean for Research, and Director of the Borish Center for Ophthalmic Research, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kollbaum002
Record Dates: First submitted 2019-02-27; First posted 2019-03-19 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hyperopia; Myopia
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lotrafilcon B (Placebo Comparator)
  Interventions: Device: Lotrafilcon B; Device: lotrafilcon B with Hydraluxe
- Lotrafilcon B Hydraluxe (Active Comparator)
  Interventions: Device: Lotrafilcon B; Device: lotrafilcon B with Hydraluxe

INTERVENTIONS:
Device: Lotrafilcon B — commercially available contact lens
Device: lotrafilcon B with Hydraluxe — commercially available contact lens

SUMMARY:
The current study aims to systematically investigate the diurnal variation in the optical quality of soft contact lenses on eye throughout the day. Subject reported quality of vision will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Habitual prescription +5.00 D to -6.00 D
* 18-35 years of age
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* Vertex corrected refractive cylinder must be -0.75 or less.
* Visual acuity best correctable to 20/25 or better for each eye
* The subject must read and sign the Informed Consent form.
* Mesopic pupil size >5.00 mm.

Exclusion Criteria:

* active condition that would prevent contact lens wear
* history of issues of eye alignment or binocularity by self-report
* doctor diagnosed, self-reported accommodative or binocular vision issues
* doctor diagnosed, self-reported ocular surface disease or dry eye requiring regular, ongoing treatment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Clinical Optics Research Lab, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotrafilcon B First, Then Lotrafilcon B With Hydraluxe; Lotrafilcon B With Hydraluxe First, Then Lotrafilcon B: First intervention (2+/-1day) Second intervention (2+/-1day)
Period: Overall Study
Arm/Group | Lotrafilcon B First, Then Lotrafilcon B With Hydraluxe | Lotrafilcon B With Hydraluxe First, Then Lotrafilcon B
Started | 12 | 12
Completed First Intervention | 12 | 12
Completed Second Intervetion | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotrafilcon B First, Then Lotrafilcon B With Hydraluxe | Lotrafilcon B With Hydraluxe First, Then Lotrafilcon B | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.25 (3.57) | 24.33 (3.80) | 24.29 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 8 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Higher Order Aberrations
Description: Higher-order Root Mean Squared (RMS) over a 3mm pupil; difference in RMS error between 0 and 12 hour timepoints; averaged across all subjects
Time Frame: 0-12 hours
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Lotrafilcon B; Lotrafilcon B With Hydraluxe: All subjects (randomized, crossover design)
Arm/Group | Lotrafilcon B | Lotrafilcon B With Hydraluxe
Number analyzed (Participants) | 24 | 24
microns | 0.001646 (0.028867) | 0.002629 (0.044299)

2. Secondary Outcome: Subjective Stability of Vision Rating
Description: Subjects are asked to rate their stability of vision on a numeric rating scale (0, poor to 100 excellent) (Kollbaum 2012). The difference between time 0 and time 12 hours is reported for all subjects (negative number represents a decrease in stability of vision)
Time Frame: 0-12 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lotrafilcon B | Lotrafilcon B Hydraluxe
Number analyzed (Participants) | 24 | 24
score on a scale | -5.833 (10.8) | -2.500 (9.78)
Statistical Analysis 1: Comparison: Lotrafilcon B; Change in ratings over time; Test type: Other — Friedman test; p = 0.0023, Friedman Test
Statistical Analysis 2: Comparison: Lotrafilcon B Hydraluxe; change in ratings over time; Test type: Other — Friedman test; p = 0.4679, Friedman Test

3. Secondary Outcome: Image Quality Metrics
Description: Root Mean Squared (RMS) wavefront error over a 3mm pupil; difference in RMS error between 0 and 12 hour timepoints; averaged across all subjects
Time Frame: 0-12 hours
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Lotrafilcon B | Lotrafilcon B With Hydraluxe
Number analyzed (Participants) | 24 | 24
microns | 0.015134 (0.051825) | 0.013899 (0.036077)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 weeks
Groups:
- Lotrafilcon B: During wear of Lotrafilcon B, including all subjects, despite randomization
- Lotrafilcon B With Hydraluxe: During wear of Lotrafilcon B With Hydraluxe, including all subjects, despite randomization
Arm/Group | Lotrafilcon B | Lotrafilcon B With Hydraluxe
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03881670/Prot_SAP_000.pdf